CLINICAL TRIAL: NCT06050629
Title: The Characteristics of Backscattering With Depth in the Progression of Keratoconus and Its Role in Forme Fruste Keratoconus Detection
Brief Title: The Characteristics of Backscattering With Depth in the Progression of Keratoconus
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2023020
Record Dates: First submitted 2023-09-08; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Elasticum, Incomplete Pseudoxanthoma
MeSH Terms: conditions — Pseudoxanthoma Elasticum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- forme fruste keratoconus: 1) no other eye abnormalities except myopia and astigmatism; 2) transparent cornea; 3) no positive signs of keratoconus on slit lamp examination or morphology examination (excluding the appearance of keratoconus as described above, and simultaneously satisfying A0B0C0D0, Index of Surface variance (ISV) < 30, and Keratoconus Index (KI) < 1.07); and 4) Belin/Ambrósio enhanced ectasia total derivation value(BAD-D)≤1.6
- Clinical keratoconus: 46.5 D ≤ Mean K <52 D; 55≤ ISV<200; and 1.10 ≤ KI <1.50
- severe keratoconus: Mean K ≥ 52D; ISV≥ 200; and KI≥ 1.50
- normal eye: one eye of healthy participants before refractive surgery were randomly selected. Comprehensive ophthalmic examinations were performed before surgery, which confirmed that the cornea was clear and normal in shape. For this group, there was no family history of keratoconus, no other diseases except ametropia, and no corneal dilatation one year after surgery.

SUMMARY:
To investigate the variation in backscattering with depth between forme fruste keratoconus (FFKC), keratoconus, and normal eyes; to determine the backscattering changes in the characteristics of keratoconus progression; and to explore the diagnostic value of backscattering in FFKC.

DETAILED DESCRIPTION:
To investigate the variation in backscattering with depth between forme fruste keratoconus (FFKC), keratoconus, and normal eyes; to determine the backscattering changes in the characteristics of keratoconus progression; and to explore the diagnostic value of backscattering in FFKC. A Scheimpflug corneal tomography image and caliper tool were used to obtain backscatter at every 2% depth at the thinnest point of the cornea, with the measured values expressed in grayscale units (GSU).

ELIGIBILITY:
Inclusion Criteria:

1. BCVA <20/20 and a history of myopia or astigmatism;
2. presence of any of the following positive signs on slit lamp examination: corneal stromal thinning, cone-shaped anterior protrusions, Fleischer's ring, Vogt's striae, epithelial or subepithelial scarring;
3. abnormal corneal topography (maximum keratometry (K) value of >47.2 diopters (D), bow-tie pattern with skewed radial axes, or inferior-superior asymmetry(3-mm I-S keratometric difference >1.4 D).

Exclusion Criteria:

1. Patients with severe corneal scarring that affected light scattering and density maps showing "black holes" 2.Participatients with other corneal diseases 3. Eyes that have undergone surgery or trauma 4. Eyes with corneal dystrophy

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study was performed on patients with keratoconus and healthy participants admitted to Tianjin Eye Hospital from January 2020 to December 2022.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
backscattering | through study completion, an average of 1 year
  Standard measurements were performed using a Pentacam (Pentacam HR; Oculus, Wetzlar, Germany);The average brightness of a predetermined area of the cornea was calculated, shown as densitometry, and recorded in GSU ranging from 0 to 100 (0, cornea is transparent without opacity; 100, cornea is completely opaque).

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided